CLINICAL TRIAL: NCT06655324
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Trial to Evaluate the Safety, Tolerability, and Immunogenicity of V350A and V350B in Healthy Participants.
Brief Title: A Study to Evaluate Safety, Tolerability, and Immunogenicity of V350A and V350B in Healthy Participants (V350-001).
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: V350-001
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- V350A (Experimental): Participants will receive V350A vaccinations on Day 1, Month 2, and Month 6.
  Interventions: Biological: V350A
- V350B (Experimental): Participants will receive V350B vaccinations on Day 1, Month 2, and Month 6.
  Interventions: Biological: V350B
- Placebo (Placebo Comparator): Participants will receive placebo vaccinations on Day 1, Month 2, and Month 6.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V350A — Vaccination administered via intramuscular injection
  Arms: V350A
Biological: V350B — Vaccination administered via intramuscular injection
  Arms: V350B
Biological: Placebo — Vaccination administered via intramuscular injection
  Arms: Placebo

SUMMARY:
Epstein Barr virus (EBV) is a virus which can cause infectious mononucleosis and is associated with certain kinds of cancer and multiple sclerosis. Researchers are looking for new ways to prevent disease related to EBV and have developed a new study vaccine (V350A and V350B). The main goal of this study is to learn about the safety and tolerability of V350A and V350B in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization.
* Has a body mass index ≥18 and ≤38 kg/m^2, inclusive.

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a confirmed or suspected case of infectious mononucleosis within 12 months prior to enrollment.
* Has any immunosuppressive medical condition or receive any immunosuppressive therapy.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2028-07-17 (Estimated); Study Completion 2028-07-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Solicited Injection Site Adverse Events (AEs) | Up to approximately 6 months
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited injection site AEs will be recorded on a vaccination report card (VRC).
Number of Participants with Solicited Systemic AEs | Up to approximately 6 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Solicited systemic AEs will be recorded on a VRC.
Number of Participants with Immediate AEs Following Vaccinations | Up to approximately 6 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Participants will be observed following vaccination for immediate AEs.
Number of Participants with Unsolicited AEs | Up to approximately 7 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Unsolicited AEs will be recorded on a VRC.
Number of Participants with Serious AEs | Up to approximately 18 months
  A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event.
Number of Participants with Medically Attended Adverse Events (MAAEs) | Up to approximately 18 months
  A MAAE is an AE in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an emergency department visit, office visit, or an urgent care visit with any medical personnel for any reason. Routine visits are not considered MAAEs.
Number of Participants with Events of Clinical Interest (ECIs) | Up to approximately 18 months
  ECIs are selected serious and nonserious AEs are defined as an overdose of Sponsor's product, drug-induced liver injury events, or potential immune-mediated diseases (pIMDs).

SECONDARY OUTCOMES:
Geometric Mean Titers (GMT) of Immunoglobulin G (IgG) Antibodies Response Against Vaccine-matched Epstein Barr Virus (EBV) Antigens | Up to approximately 18 months
  The GMT of EBV antigen antibody titers will be measured with a multiplex ligand binding assay (LBA).
Geometric Mean Fold Rise (GMFR) of IgG Antibody Response against Vaccine-matched EBV Antigens | Baseline and up to approximately 18 months
  The GMFR of EBV antigen antibody titers will be measured with a multiplex LBA.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- United States (9):
  - California Clinical Trials Medical Group managed by PAREXEL ( Site 0011), Glendale, California
  - QPS-MRA, LLC ( Site 0012), Miami, Florida
  - Alliance for Multispecialty Research, LLC ( Site 0008), Kansas City, Missouri
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO ( Site 0016), Springfield, Missouri
  - Velocity Clinical Research Lincoln ( Site 0004), Lincoln, Nebraska
  - Velocity Clinical Research, Omaha ( Site 0005), Omaha, Nebraska
  - Remington-Davis, Inc. ( Site 0017), Columbus, Ohio
  - Lynn Health Science Institute ( Site 0010), Oklahoma City, Oklahoma
  - Alliance for Multispecialty Research, LLC ( Site 0009), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com